CLINICAL TRIAL: NCT00672490
Title: An Open Label, 4-Week, Randomised, Multi-Centre, Phase IV Study to Compare the Efficacy and Safety of Quetiapine Fumarate (Seroquel) as Mono-Therapy or Adjunct to Lithium in the Treatment of Patients With Acute Mania in Bipolar Disorder
Brief Title: Quetiapine Fumarate (Seroquel) as Mono-Therapy or Adjunct to Lithium in the Treatment of Patients With Acute Mania in Bipolar Disorder
Acronym: MANIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00023
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Acute Mania in Bipolar Disorder
Keywords: Acute Mania; Bipolar Disorder; Quetiapine Fumarate; Lithium
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quetiapine Fumarate - tablets
  Interventions: Drug: Quetiapine Fumarate
- 2 (Experimental): Quetiapine Fumarate - tablets and Lithium
  Interventions: Drug: Quetiapine Fumarate; Drug: Lithium

INTERVENTIONS:
Drug: Quetiapine Fumarate — Oral treatment, twice daily. 100 mg/day at Day 1, 200 mg/day at Day 2, 300 mg/day at Day 3, 400 mg/day at Day 4, from 400 mg/day to 600 mg/day before Day 8, from 600 mg/day to 800 thereafter, judged by the investigator.
  Tablets
  Other Names: Seroquel
Drug: Lithium — Oral treatment, twice daily. 250 mg/day to 2000mg/day from Day1 to Day 7, 500mg/day to 2000mg/day thereafter, judged by the investigator.
  Arms: 2

SUMMARY:
To compare the efficacy and safety of quetiapine fumarate given as mono-therapy or adjunct therapy to lithium in the treatment of patients with acute mania in bipolar disorder. Patients with a documented clinical diagnosis of bipolar mania according to DSM-IV criteria (296.4X Bipolar I Disorder, Most Recent Episode Manic; 296.0X Bipolar I Disorder, Single Manic Episode) are required to have a YMRS total score of ≥20 at enrolment and randomisation

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent before initiation of any study related procedures. Patients who are deemed incapable of providing informed consent maybe enrolled if written informed consent has been obtained from the patient's Legally Authorized Representative.
* Documented clinical diagnosis meeting the DSM-IV criteria for any of the following:
* 296.4X Bipolar I Disorder, Most Recent Episode Manic
* 296.0X Bipolar I Disorder, Single Manic Episode
* Have a YMRS score of at least 20 and a score of at least 4 on 2 of the following 4 YMRS items both at enrolment and at randomisation: Irritability, Speech, Content, and Disruptive/Aggressive Behaviour.
* Female patients of childbearing potential must have a negative urine pregnancy test at enrolment and be willing to use a reliable method of birth control, i.e., barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation, during the study.
* Be able to understand and comply with the requirements of the study, as judged by the investigator.

Exclusion Criteria:

* Manic episode judged to be either:
* the direct physiological consequence of a treatment or medical condition other than Bipolar disorder.
* the direct physiological effect of a substance of abuse; intoxication with hallucinogens, inhalants, opioids, or phencyclidine and related substances.
* the direct physiological effect of psychostimulant or antidepressant medication.
* Evidence of clinically severe or active disease, or a clinical finding that is unstable or that, in the opinion of the investigator, would be negatively affected by the study medication or that would affect the study medication.
* History of seizure disorder, except febrile convulsions.
* Hospitalization period of 3 weeks or longer immediately prior to randomization for the index manic episode.
* Known history of intolerance or hypersensitivity to quetiapine or lithium, or to any other component in the tablets/capsules.
* Known lack of response to quetiapine or lithium, as judged by the investigator.
* Use of antipsychotic medication or mood stabilizer other than quetiapine and lithium at the day of randomisation (to be tapered to discontinuation between the enrolment visit and randomisation).
* Administration of a depot antipsychotic injection within 1 dosing interval (for the depot) before randomisation.
* Use of clozapine within 28 days prior to randomisation.
* Use of antidepressants during the enrolment period or within a period of 5 half-lives of the drug(s) prior to randomisation.
* Continuous daily use of benzodiazepines in excess of 4 mg per day of lorazepam, or the equivalent, during 28 days prior to randomisation.
* Use of drugs that induce or inhibit the hepatic metabolizing cytochrome 3A4 enzymes within 14 days before randomisation.
* Receipt of electroconvulsive therapy (ECT) within 28 days prior to randomisation.
* Clinically significant deviation from the reference range in clinical laboratory test results at enrolment, as judged by the investigator.
* An absolute neutrophil count (ANC) of <1.5X109/L.
* Treatment with quetiapine with a dosage of at least 50 mg/day at enrolment (Visit 1)
* Liver function test AST or ALT 2 times as the upper normal limit.
* A thyroid-stimulating hormone (TSH) concentration more than 10% above the upper limit of the normal range of the laboratory used for sample analysis at enrolment, whether or not the subject is being treated for hypothyroidism.
* Known diagnosis of Diabetes Mellitus (DM) or fasting blood glucose level > the upper normal limit.
* Risk of transmitting human immuno-deficiency virus (HIV) or hepatitis B via blood or other body fluids, as judged by the investigator.
* ECG results considered to be clinically significant as determined by the investigator.
* Conditions that could affect absorption and metabolism of study medication.
* Patients who in the investigators opinion will require systematic psychotherapy (other than supportive psychotherapy) during the study period.
* Participation in another clinical study or compassionate use programme within 28 days prior to randomisation, or longer if locally required.
* Involvement in the planning and conduct of the study (applies to all AstraZeneca or staff at the investigational site).
* Previous enrolment or randomisation of treatment in the present study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 376 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Hongyan, Prof., Principal Investigator — Peking University 6th hospital
Locations (16):
- China (16):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Baoding, Hebei
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Daqing, Heilongjiang
  - Research Site, Xinxiang, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Suzhou, Jiangsu
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xijing, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kuming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Huzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine Fumarate Used as Mono-Therapy: Quetiapine Fumarate 600 to 800 mg/day
- Quetiapine Fumarate Used as Adjunct Therapy: Quetiapine Fumarate 600 to 800 mg/day + lithium 500 mg to 2000 mg/day
Period: Overall Study
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Started | 187 | 189
Completed | 163 | 157
Not Completed | 24 | 32
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Lack of Compliance | 2 | 7
Not completed — Mismatch Include/Exclude Criteria | 1 | 0
Not completed — Adverse Event | 5 | 8
Not completed — Violation of Concomitant Medicine | 1 | 0
Not completed — Intolerance | 0 | 2
Not completed — Lost to Follow-up | 1 | 5
Not completed — No reason was provided | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy | Total
Number analyzed (Participants) | 187 | 189 | 376
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.16) | 32.43 (11.14) | 33.36 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 87 | 181
  Male | 93 | 102 | 195

OUTCOME MEASURES:

1. Primary Outcome: Change in the Young Mania Rating Scale (YMRS) Total Score From Baseline to Final Assessment (Day 28)
Description: The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).
Time Frame: Baseline and 4 weeks
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 178 | 178
score on a scale | -25.7 (13.7) | -26.1 (13.4)

2. Secondary Outcome: Change From Baseline in the Clinical Global Impressions for Bipolar Disorder Severity of Illness (CGI-BP-S) Score to Each Assessment (Day 28)
Description: The CGI-BP-S scale rates the severity of the patient's illness at the time of assessment and is scored from 1 to 7 (1=normal, not ill to 7=very severely ill). Higher CGI-BP-S scores indicate greater illness severity
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
score on a scale | -2.65 (0.115) | -0.17 (0.144)

3. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score to Each Assessment (Day 28)
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia and each item is rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 individual-item scores and ranges from 30 to 210
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
units on a scale | -16.12 (0.285) | -16.44 (0.28)

4. Secondary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score to Each Assessment(Day 28)
Description: The MADRS is a 10-item scale that evaluates depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. Higher MADRS scores indicate higher levels of depressive symptoms. The MADRS total score is the sum of all 10 individual-item scores and ranges from 0 to 60.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
score on a scale | -2.99 (0.181) | -3.02 (0.179)

5. Secondary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) Item 4 Score to Each Assessment
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 4 (sleep) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
score on a scale | -2.0 (1.2) | -2.1 (1.2)

6. Secondary Outcome: Response Rate (Number of Patients With Clinically Response)
Description: The number of patients with clinically response (defined as ≥50% reduction in the YMRS total score from baseline to Day 28) was calculated. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or 50% reduction) from baseline indicates a reduction (or improvement) in manic symptoms.
Time Frame: From Baseline to 4 weeks
Measure: Number; unit: Participants
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
Participants | 139 | 153

7. Secondary Outcome: Remission Rate (Number of Patients With Clinically Significant Remission)
Description: The number of patients with clinically significant remission (defined as YMRS total score ≤12) at Day 28 was calculated.
  The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania. Total score ≤12 indicates remission.
Time Frame: From Baseline to 4 weeks
Measure: Number; unit: Participants
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
Participants | 117 | 123

8. Secondary Outcome: Treatment of Agitation (Change From Baseline in the PANSS Activation Subscale Score to Day 28)
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia and each item is rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS activation subscale score for effect on agitation and aggression is the sum of 6 PANSS individual items (ie, hostility, poor impulse control, excitement, uncooperativeness, poor rapport and tension) and ranges from 6 to 42.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
score on a scale | -5.4 (4.5) | -5.8 (4.2)

9. Secondary Outcome: Treatment of Aggression Risk (Change From Baseline in the PANSS Supplement Aggression Risk Subscale Score to Day 28)
Description: The PANSS Supplemental Aggression Risk subscale score is the sum of 3 standard PANSS items - Excitement, Hostility and Depression - and 3 supplemental PANSS items related to anger - Anger, Difficulty in Delaying Gratification and Affective Lability and ranges from 6 to 42, where 6 is the "best" and 42 the "worst" score for the combined scale.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Number analyzed (Participants) | 187 | 189
score on a scale | -6.8 (5.1) | -7.3 (5.1)

ADVERSE EVENTS:
Arm/Group | Quetiapine Fumarate Used as Mono-Therapy | Quetiapine Fumarate Used as Adjunct Therapy
Serious Adverse Events (participants affected / at risk) | 0/187 | 1/189
Other Adverse Events (participants affected / at risk) | 120/187 | 125/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine Fumarate Used as Mono-Therapy (N=187) | Quetiapine Fumarate Used as Adjunct Therapy (N=189)
Injury (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine Fumarate Used as Mono-Therapy (N=187) | Quetiapine Fumarate Used as Adjunct Therapy (N=189)
Constipation (Gastrointestinal disorders) | 13 | 24
Nausea (Gastrointestinal disorders) | 4 | 15
Vomiting (Gastrointestinal disorders) | 1 | 10
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Weight Increased (Investigations) | 12 | 16
Dizziness (Nervous system disorders) | 21 | 14
Extrapyramidal Symptom (Nervous system disorders) | 6 | 12
Somnolence (Nervous system disorders) | 10 | 10
Tremor (Nervous system disorders) | 5 | 13
Tachycardia (Cardiac disorders) | 11 | 7
Palpitations (Cardiac disorders) | 7 | 4
Hypothyroidism (Endocrine disorders) | 0 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 9
Dry mouth (Gastrointestinal disorders) | 3 | 6
Fatigue (General disorders) | 4 | 6
Liver function test abnormal (Investigations) | 8 | 9
Hyperlipidemia (Metabolism and nutrition disorders) | 3 | 7
Hypersomnia (Nervous system disorders) | 13 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other